CLINICAL TRIAL: NCT04938921
Title: Short-term and Mid-term Outcome of Sutureless Closure for Primary Total Anomalous Pulmonary Venous Connection
Brief Title: Sutureless Closure for Primary Total Anomalous Pulmonary Venous Connection
Acronym: TAPVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital 1 (Other)
Responsible Party: Principal Investigator, Thanh QL. Dinh, MD, Ms, Principle investigator, Children's Hospital 1
Other Study IDs: 3685/QD-DHYD
Record Dates: First submitted 2021-06-16; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Total Anomalous Pulmonary Venous Connection; Pulmonary Venous Stenosis; Sutureless Closure
Keywords: TAPVC; Sutureless; Pulmonary venous stenosis
MeSH Terms: conditions — Scimitar Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the percentage of pulmonary venous stenosis after TAPVC repair with sutureless closure.

DETAILED DESCRIPTION:
Parents of patients with TAPVC after repairing by sutureless technique will be informed about the study. If parents agree to participant in the study and sign the informed consent, the investigators will collect information of patients and echocardiography results at 1 month, 6 month, 12 month and 18 month after the operation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with TAPVC operated with sutureless closure and be agreed to join this study by parents from 01/2019 to 06/2024.

Exclusion Criteria:

* TAPVC operated with sutureless closure have single ventricle, isomerism or heterotaxy, congenital pulmonary venous stenosis.
* TAPVC enrolled to study but cannot the obtain the echocardiography at the time of 1 month, 6 month, 12 month and 18 month.

Max Age: 15 Years | Sex: All
Age Groups: Child
Study Population: All patients with TAPVC operated with sutureless closure and be agreed to joint this study by parents from 01/2019 to 06/2024
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of pulmonary venous stenosis after reparing TAPVC with sutureless technique | The investigators assess the PVS at the time of 12 month after the operation.
  The investigators calculate pulmonary venous score (PVS) based on the mean gradient through each pulmonary vein. Then we sum all the score of each pulmonary vein, range from 0 to 12, and classify to 4 levels. Score 0 if the mean gradient is less than 2mmHg, 1 if it is from 2 to 6,9mmHg, 2 if it is from 7 mmHg and above, and 3 if the vein is occluded. The degree of obstruction is classified as follow: none (0 to 1), mild (2 to 3), moderate (4 to 7), and severe (from 8 and above).
Early mortality (<30 days) | 30 days
  Early mortality is defined when patients die within 30 days since the operation
The percentage of pulmonary venous stenosis after reparing TAPVC with sutureless technique | The investigators assess the PVS at the time of 18 month after the operation.
  The investigator calculate pulmonary venous score (PVS) based on the mean gradient through each pulmonary vein. Then we sum all the score of each pulmonary vein, range from 0 to 12, and classify to 4 levels. Score 0 if the mean gradient is less than 2mmHg, 1 if it is from 2 to 6,9mmHg, 2 if it is from 7 mmHg and above, and 3 if the vein is occluded. The degree of obstruction is classified as follow: none (0 to 1), mild (2 to 3), moderate (4 to 7), and severe (from 8 and above).

SECONDARY OUTCOMES:
Late mortality (> 30 days) | The investigators assess mortality at the time of 18 month after the operation
  Late mortality is defined when patients die beyond 30 day since the operation
The percentage of pulmonary venous stenosis after reparing TAPVC with sutureless technique | The investigators assess the PVS at the time of 6 month after the operation.
  The investigator calculate pulmonary venous score (PVS) based on the mean gradient through each pulmonary vein. Then we sum all the score of each pulmonary vein, range from 0 to 12, and classify to 4 levels. Score 0 if the mean gradient is less than 2mmHg, 1 if it is from 2 to 6,9mmHg, 2 if it is from 7 mmHg and above, and 3 if the vein is occluded. The degree of obstruction is classified as follow: none (0 to 1), mild (2 to 3), moderate (4 to 7), and severe (from 8 and above).

CONTACTS AND LOCATIONS:
Overall Officials: Thoi K Ngo, MSC, Study Director — Children's Hospital 1; Phuc M Vu, PhD, Study Director — University of Medicine and Pharmacy in HCMC; Tuan D Nguyen, MSC, Study Director — Children's Hospital 1; Linh NU Truong, PhD, Study Director — University of Medicine and Pharmacy in HCMC
Locations (1):
- Children's Hospital 1, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided